CLINICAL TRIAL: NCT03457246
Title: Efficacy and Tolerance of D-pigment Versus Moisturizer in Hands' Lentigo Lesions With or Without Laser Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RV4280A2012607
Record Dates: First submitted 2018-02-14; First posted 2018-03-07 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-02

CONDITIONS: Lentigo; Hyperpigmentation
Keywords: solar lentigos; physical Hyperpigmentation therapies; cosmetic topical depigmenting product; topical Hyperpigmentation therapies
MeSH Terms: conditions — Lentigo; Hyperpigmentation

STUDY DESIGN:
Intervention Model Description: intra-individual hand controlled trial (left/ right comparison)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- D-Pigment rich texture (Experimental): Hand with 5 to 10 lentigos (graded 6 or more on the severity grading scale) treated by test product ( D-pigment rich texture).
  Interventions: Other: D-Pigment rich texture
- Hydrance optimale riche (Placebo Comparator): Hand with 5 to 10 lentigos (graded 6 or more on the severity grading scale) treated by reference product (Hydrance optimale riche)
  Interventions: Other: Hydrance optimale riche

INTERVENTIONS:
Other: D-Pigment rich texture
  Other Names: Dermo-cosmetic product
  Arms: D-Pigment rich texture
Other: Hydrance optimale riche
  Other Names: Dermo-cosmetic product
  Arms: Hydrance optimale riche

SUMMARY:
Pierre Fabre Dermo-Cosmétique has commercialized a cosmetic product (D-pigment rich texture) for treatment of hyperpigmentation. The aim of this study is to evaluate the efficacy of D-pigment after laser therapy, through its action on peri-lesional areas, in obtaining better cosmetic effect.

DETAILED DESCRIPTION:
Many studies have shown the efficacy of topical products such as hydroquinone, tretinoin, ascorbic and phytic acid... The combination of topical agents has shown better improvement of lentigos aspect. Many physical therapy such as chemical peels, cryosurgery, dermabrasion, and pigment-specific lasers show good results.

The combination of physical and topical therapies may be beneficial to patients. For example, the use of combination topical therapy may be used after cryotherapy as a maintenance therapy to diminish the risk of relapse. Laser therapy is very efficient on visible lesion, but not to prevent lesions apparition. A cosmetic topical depigmenting product may be a support of laser therapy, to prevent lentigos apparition in peri-lesional areas.

Furthermore, Post-inflammatory hyperpigmentation (PIH) is a common adverse effect seen with laser, occurring in approximately 35-40% of patients with Fitzpatrick skin types I-III. Another study related that 28% of study population has post-inflammatory hyperpigmentation. A cosmetic topical depigmenting product may be a support of laser therapy, to prevent possible laser side effect.

Pierre Fabre Dermo-Cosmétique has commercialized a cosmetic product (D-pigment rich texture) for treatment of hyperpigmentation. The aim of this study is to evaluate the efficacy of D-pigment as a support of a laser therapy, through its action on peri-lesional areas.

The expected effect is to show the efficacy of D-pigment in post laser long-term treatment, having a more homogenous skin colour on the D-pigment hand versus the moisturizer hand. The subjects will benefit from a strengthened follow-up by the investigator (one visit every 3 months). After the completion of the study, a complete hands laser treatment will be done for each subject and D-pigment tubes will be offered to the subjects for a 6 months application period.

ELIGIBILITY:
Inclusion Criteria:

* Subject consenting on the use of photos for scientific and commercial purposes,
* Subject having signed his/her written informed consent.
* Subject treated by laser therapy in the previous 15 to 30 days
* Subject having 5 to 10 lentigos on the surface of each hands
* Subject having lentigos graded 6 or more on the severity grading scale
* Subject with same lentigo severity in each hand.

Exclusion Criteria:

* Subject who has planned to stay for more than 15 days in an area with an important increase in sun exposure conditions compared to his/her usual place of residence,
* Subject who has planned to sun expose himself/herself more than 7 days,
* Women with childbearing potential
* Participation to an other clinical trial in the previous month or during the study,
* Subject who is not able to understand the information (for linguistic or psychiatric reasons), to give informed consent,
* Subject who, in the judgement of the investigator, is not likely to be compliant with study-related constraints during the study (daily product application during one year),
* Subject who has forfeited her freedom by administrative or legal decision, or who is under guardianship.

Criteria related to pathologies:

* Hyperpigmentation other than lentigos or other hypermelanosis (post-inflammatory laser or chemical melanosis) on the hands,
* Diabetic subject,
* Chronic or progressive disease which may interfere with the study in the opinion of the investigator,
* Pathology, skin disorder or lesions other than lentigo (psoriasis, atopic dermatitis, mycose, intertrigo, sunburn…) at the dorsum of the hand which could interfere with the evaluation,
* Systemic infectious pathology,
* Hypersensitivity, allergy or intolerance to retinaldehyde or any component of the formulation.

Criteria related to treatments:

* Treatment by depigmenting cosmetic products on the hands within 4 weeks prior to inclusion,
* Treatment by depigmenting treatment containing hydroquinone or any depigmenting drug on the hands (e.g. topical retinoids, topical steroids, …) within 8 weeks prior to inclusion,
* Previous treatment by chemical peels, dermabrasions on the hands within one year prior to inclusion,
* Treatment by photosensitive agents within 8 weeks prior to inclusion.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-05-06 (Actual); Primary Completion 2014-06-10 (Actual); Study Completion 2014-06-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline skin color homogeneity at 12 months by blinded evaluation from standardized photos. | Assessed at 12 months versus baseline.
  Scoring homogeneity will be assessed through 2 Visual Analogue Scales. One VAS grades the surface affected by lentigo on observed area, no lentigo corresponding to 0 and area completely hidden by lentigo to 10.
  The second VAS grades differences between lighter and darker skin of areas, same color skin corresponding to 0 and extremely dark lentigo to 10.
  Sum of the two VAS (0 to 20) represents the homogeneity of the skin color Blinded evaluation.
  During all the visits, an investigator will take photos. After visits, photos will be renamed and resampled. The investigator who will evaluate the parameter may be independent from that one who took photos.
  Each parameter will be evaluated by the same person avoiding thus quotation bias. They will be evaluated on each area blinded from product applied and from time evaluated.
  The appraiser will quote at the same time the pictures obtained for one subject, for one hand, at Baseline and at 12 months.

SECONDARY OUTCOMES:
Change over time of skin color homogeneity by blinded evaluation from standardized photos. | assessed at Day 0, 3 months, 6 months, and 9 months.
  Scoring homogeneity will be assessed through 2 Visual Analogue Scales. One VAS grades the surface affected by lentigo on observed area, no lentigo corresponding to 0 and area completely hidden by lentigo to 10.
  The second VAS grades differences between lighter and darker skin of areas, same color skin corresponding to 0 and extremely dark lentigo to 10.
  Sum of the two VAS (0 to 20) represents the homogeneity of the skin color Blinded evaluation.
  During all the visits, an investigator will take photos. After visits, photos will be renamed and resampled. The investigator who will evaluate the parameter may be independent from that one who took photos.
  Each parameter will be evaluated by the same person avoiding thus quotation bias. They will be evaluated on each area blinded from product applied and from time evaluated.
  The appraiser will quote at the same time the pictures obtained for one subject, for one hand, at the different times evaluated for the study.
Change over time of skin color homogeneity by clinical evaluation. | assessed at Day 0, 3 months, 6 months, 9 months and 12 months.
  An Investigator will grade the skin colour homogeneity by clinical evaluation through 2 Visual Analogue Scales.
  One VAS grades the surface affected by lentigo on observed area, no lentigo corresponding to 0 and area completely hidden by lentigo to 10.
  The second VAS grades differences between lighter and darker skin of areas, same color skin corresponding to 0 and extremely dark lentigo to 10.
  Sum of the two VAS (0 to 20) represents the homogeneity of the skin color.
Lentigos number by clinical evaluation | assessed at Day 0, 3 months, 6 months, 9 months and 12 months
  At each visit the investigator will examine the subject, count the number of lentigos and report the number on the CRF.
Lentigos number by blinded count from standardized photos. | assessed at Day 0, 3 months, 6 months, 9 months and 12 months
  During all the visits, an investigator will take photos. After visits, photos will be renamed and resampled. The investigator who will count the number of lentigos may be independent from that one who took photos.
  The count will be performed by the same person avoiding thus quotation bias. Lentigos will be count on each area blinded from product applied and from time evaluated.
  The appraiser will quote at the same time the pictures obtained for one subject, for one hand, at the different times evaluated for the study.
Evaluation of lentigo Color versus healthy surrounding skin color by Colorimetry (L*, a*, b*) | assessed at Day 0, 3 months, 6 months, 9 months and 12 months
  Colorimetric measurements of the coloration are performed by a colorimeter. Skin color is characterized according to 3 components of the three-dimensional colorimetric space L *, a *, b *, where L* represents the brightness ( black / white axis), a* represent the redness ( green / red axis), b* represent the 'yellow' ( blue / yellow axis).
  Four lentigos as "target lesions" will be selected. Colorimetric measurements will be performed on each and compared to those of healthy surrounding skin.
Pigment distribution of lentigos assessed by In vivo Reflectance Confocal Microscopy (RCM) | assessed at Day 0, 3 months, 6 months, 9 months and 12 months
  Four lentigos as "target lesions" will be selected and imaged by RCM :
  Pigment distribution will be evaluated through a 5 points scale. 0 = Absence of pigment on the study area
  1. < 10 %,
  2. = between 10-30%,
  3. = between 30-50%,
  4. > 50% of the study area covered by pigment
Enlarged interpapillary spaces of lentigos assessed by In vivo Reflectance Confocal Microscopy (RCM) | assessed at Day 0, 3 months, 6 months, 9 months and 12 months
  Four lentigos as "target lesions" will be selected and imaged by RCM. Interpapillary spaces will be evaluated through a 4 points scale. 0 = Absence of interpapillary space
  1. < 10 %,
  2. = between 10-30%,
  3. = interpapillary space is between 30-50% of papillary size
Intensity of papillary brightness of lentigos assessed by In vivo Reflectance Confocal Microscopy (RCM) | assessed at Day 0, 3 months, 6 months, 9 months and 12 months
  Four lentigos as "target lesions" will be selected and imaged by RCM. Interpapillary spaces will be evaluated through a 3 points scale.
  1= low brightness 2 = medium 3= hight brightness
Signs of inflammation in lentigos assessed by In vivo Reflectance Confocal Microscopy (RCM) | assessed at Day 0, 3 months, 6 months, 9 months and 12 months
  Four lentigos as "target lesions" will be selected and imaged by RCM. inflammation signs will be evaluated through a 3 points scale. 0 = Absence of inflammation signs
  1. < 10 %,
  2. = between 10-30% of the study area covered by inflammation signs
Dynamic Physician Global Assessment (PGA) | assessed at 3 months, 6 months, 9 months and 12 months
  For this parameter, four "target lesions" will be selected for the analysis: one previous treated by laser and one not treated by laser on each hand. The instrument's field of view will allow exploring parameters on the target lesions and the peri-lesional area.
Overall efficacy assessed by the Subject | assessed at 3 months and 12 months
  The overall efficacy is defined through a 5 points scale. 0 = completely improved
  1. = mostly improved
  2. = slightly improved
  3. = no improvement
  4. = worse
  The subjects will assess the overall efficacy on each global hand, on area treated by laser and area not treated by laser of each hand.
  The efficacy assessed by the subjects will be compared at 3 and 12 months of product application between :
  * D-pigment hand versus moisturizer hand
  * area treated by laser on D-pigment hand versus area treated by laser on moisturizer hand
  * area not treated by laser on D-pigment versus area not treated by laser on moisturizer hand
Satisfaction regarding to the use of D-Pigment | assessed after 3 months of daily applications
  The satisfaction regarding to the use of D-pigment (conditions of use, organoleptic properties, effects...) will be assessed by the subject through a questionnaire The overall satisfaction will be assessed by the Subject through a 5 points scale.
  1. = Much pleased
  2. = Pleased
  3. = Fairly pleased
  4. = Unpleased
  5. = Much Unpleased

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni PELLACANI, Principal Investigator — Department of Dermatology - University of Modena and Reggio Emilia

IPD SHARING:
Plan to Share IPD: No